CLINICAL TRIAL: NCT03119792
Title: Salud Integral Colombia (SI! Colombia II).
Brief Title: Salud Integral Colombia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Collaborators: Fundación Cardioinfantil Instituto de Cardiología (Other); Fundación Mario Santo Domingo (Unknown); Mobilizarte Social (Unknown); SHE Foundation (Other)
Responsible Party: Principal Investigator, Valentin Fuster, Mount Sinai Heart Director, Icahn School of Medicine at Mount Sinai
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: GCO 16-1354
Record Dates: First submitted 2017-03-21; First posted 2017-04-19 (Actual); Last update posted 2019-03-25 (Actual); Status verified 2019-03

CONDITIONS: Cardiovascular Health
Keywords: Behavioral Modification; Health Community; Community Intervention; Prevention; Cardiovascular Health; Education Intervention; Colombia
MeSH Terms: interventions — Early Intervention, Educational

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Investigational (Experimental): An education intervention will be implemented for 600 children from the original cohort (300) and comparable cohort (300) over a four month period at community centers. These sessions will occur twice a month on the weekends. The education intervention will help increase the children's knowledge of attitudes, and habits of healthy lifestyles.
  Interventions: Other: Education Intervention
- Control (Active Comparator): The control group will consist of 600 children from the original cohort (300) and comparable cohort (300). The control group will meet twice a month for four months at community centers. During these sessions, investigators will teach a curriculum that is not related to knowledge, attitudes, and habits towards healthy lifestyles.
  Interventions: Other: Control

INTERVENTIONS:
Other: Education Intervention — The education intervention will help increase the children's knowledge of attitudes, and habits of healthy lifestyles. The program will cover self care of the body and heart, emotional management, healthy diet, and physical activity.
  Arms: Investigational
Other: Control — The control will not receive an education program relating to knowledge, attitudes, nor habits of healthy lifestyles. Instead, these sessions will occur twice a month, and will last an hour and forty-five minutes. The control program is titled "Life's Challenges", which will focus on helping children develop skills necessary for day to day life, is divided into four modules: Person, Family, School, and Environment. There will be four different types of activities used throughout the program including: "Lets Think," "Lets Experiment," "We will finish with...or synthesis," and "Not here."
  Arms: Control

SUMMARY:
In May 2009 in Bogota, Colombia, the Si! program conducted a cluster randomized trial in 1216 children between the ages of 3 and 6 years old, and 928 parents with the aim of evaluating a five month education intervention to change knowledge, attitudes and habits related to a healthy diet and active lifestyle in preschoolers. The results showed that the program was feasible and effective. The Si! Program will perform a new follow up of its original children cohort, now between the ages of 9 and 13 years. The original cohort will be compared to a new comparable cohort to assess baseline knowledge, attitudes and habits of healthy lifestyles in knowledge, attitudes, habits and emotions towards a healthy lifestyles . A community pedagogical intervention in healthy lifestyles on cardiovascular health will be implemented in the intervention group.

DETAILED DESCRIPTION:
Cardiovascular disease (CVD) is a leading cause of mortality worldwide. Negative health behaviors initiated in childhood that persist through adulthood can be risk factors that predict CVD. In Colombia, poor lifestyle factors affecting childhood are very prevalent: 50% live a sedentary lifestyle, 48% have high fat and carbohydrate consumption, 30% are exposed to passive smoking, 14% are overweight or obese, 15.8% have hypercholesteremia, and 5% have hypertension.

Negative health behaviors initiated in childhood that persist through adulthood can be risk factors that predict CVD. In Colombia, poor lifestyle factors affecting childhood are very prevalent: 50% live a sedentary lifestyle, 48% have high fat and carbohydrate consumption, 30% are exposed to passive smoking, 14% are overweight or obese, 15.8% have hypercholesterolemia, and 5% have hypertension. In May 2009, in Bogota, Colombia, was conducted a cluster randomized trial (kindergartens) in 1216 children between 3 and 6 years old, and 928 parents with the aim of evaluate a five months educational intervention to change knowledge, attitudes and habits related to a healthy diet and active lifestyle in preschoolers. The results showed that the intervention was feasible and effective . Finally every 1216 children "cohort Usaquén" received the intervention, performing a follow-up at 18 and 36 months showing that the changes persisted over time

In 2016 the SI! Program will perform a new follow up of this cohort, in children between 9 and 13 years old, and under the assumption that the effects of this intervention have decreased, the researchers plan to evaluate through a randomized control trial the impact of a four months community educational intervention, in the cardiovascular health of these children and in knowledge, attitudes, habits and emotions towards a healthy lifestyle. The study will include children from the Usaquen´s cohort who are contacted and children of a comparable cohort (n = 1200), in order to achieve sustainable changes in the cardiovascular health of children, that impact the burden of disease in their adulthood.

Due to the high rate of migration within the country, given the social and economic difficulties faced by many Colombians, in 2015 the study population was scattered from 1 to 15 localities and from 14 kindergartens to more than 200 public and private schools, mostly in the Usaquen´s locality, with great variability ranging from the facilities, resources, length of the school day, number of children in each classroom, to the training of teachers and their low motivation and availability time to perform any initiative (data obtained from focus groups conducted in schools). For these reasons, it is not feasible to carry out a second educational intervention in schools. However, the investigators believe that a community-based intervention is an excellent choice for tracking this population.

The objective of this project is two-fold. First, it is to assess differences at baseline in healthy lifestyles between children from Usaquen's cohort and a comparable cohort. The study will also assess differences at baseline in cardiovascular health between parents from Usaquen's cohort, and a comparable cohort. Second, it is to assess the impact of a community pedagogical intervention in healthy lifestyles in children nine to thirteen years old.

ELIGIBILITY:
Inclusion Criteria:

* Children 9-13 years old from the original Usaquen's cohort
* Children 9-13 years old who are not included in the original cohort (comparable cohort)
* Parents of participating children

Exclusion Criteria:

* Participant unable to consent
* Parents of non-participating children
* Siblings of the Original Usaquen cohort's children that do not belong to the original cohort

Ages: 9 Years to 13 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 1216 (Actual)
Dates: Start 2016-11; Primary Completion 2018-02-13 (Actual); Study Completion 2018-02-13 (Actual)

PRIMARY OUTCOMES:
Change in Ideal Cardiovascular Health Score (ICH) | Baseline and 6 months
  Using the metrics and criteria for individual ideal health factors and behaviors, the ideal cardiovascular health score (ICH) will be calculated for each metric (poor=0, intermediate=1, ideal=2 points; range=0-14 points for all seven metrics) and categorized them into three groups: poor (0-4 points), intermediate (5-9 points), and ideal (10-14 points). Higher values represent a better outcome.
Change in KAH score in Children of the Original and Comparable Cohort | Baseline and 6 months
  Mean and standard deviation of the score of knowledge, attitudes, habits and emotions towards a healthy lifestyle in children will be determined, calculating the difference found between the baseline measurement and the measurement at the end of the study in intervened and control groups in the Original and comparable cohort. Possible differences between changes in means will be assessed using test t-test. Multi-variable models will be performed to adjust for potential con-founders.

SECONDARY OUTCOMES:
Change in ICH score in Children of the Original and Comparable Cohort | Baseline and 6 months
  Mean difference in scores and standard deviations in cardiovascular health (ICH) at the end of the study between intervened children in the Usaquen´s cohort and intervened children in the comparable cohort, will be determined, using a t-test. Multivariable models will be performed to adjust for potential confounders. The prevalence (CI 95%) of each of the 7 components of cardiovascular health rated as poor (risk factor) will be determined, calculating the difference found between the baseline measurement and the measurement at the end of the study in intervened children in the Usaquen´s cohort and intervened children in the comparable cohort. Possible differences between changes in prevalences will be evaluated using the chi-squared test.
Change in KAH score in Children of the Usaquen Cohort and Comparable Cohort | Baseline and 6 months
  Mean and standard deviation of the score of knowledge, attitudes, habits and emotions towards a healthy lifestyle will be determined, calculating the difference found between the baseline measurement and the measurement at the end of the study in intervened children in the Usaquen´s cohort and intervened children in the comparable cohort. Multivariable models will be performed to adjust for potential confounders. Possible differences between changes in means will be assessed using a t-test.
Change in ICH score in Parents of the Original and Comparable Cohort | Baseline and 6 months
  In parents, mean difference in scores and standard deviations in cardiovascular health (ICH) at the end of the study between intervened and control groups will be determined, using a t-test, differentiating between parents in the Usaquén´s cohort and a comparable cohort. Multivariable models will be performed to adjust for potential confounders. The prevalence (CI 95%) of each of the 7 components of cardiovascular health rated as poor (risk factor) will be determined, calculating the difference found between the baseline measurement and the measurement at the end of the study in intervened and control groups differentiating between parents in the Usaquén´s cohort and a comparable cohort. Possible differences between changes in prevalences will be evaluated using the chi-square test.

CONTACTS AND LOCATIONS:
Overall Officials: Valentin Fuster, MD, PhD, Principal Investigator — Icahn School of Medicine at Mount Sinai; Jorge Baxter, PhD, Study Chair — Mobilizarte Social; Jaime Cespedes, MD, Study Director — Fundación CardioInfantil de Cardiologia
Locations (1):
- Fundacion Cardioinfantil Instituto de Cardiologia, Bogotá, Colombia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Fernandez-Jimenez R, Briceno G, Cespedes J, Vargas S, Guijarro J, Baxter J, Hunn M, Santos-Beneit G, Rodriguez C, Cespedes MP, Bagiella E, Moreno Z, Carvajal I, Fuster V. Sustainability of and Adherence to Preschool Health Promotion Among Children 9 to 13 Years Old. J Am Coll Cardiol. 2020 Apr 7;75(13):1565-1578. doi: 10.1016/j.jacc.2020.01.051. PMID 32241373